CLINICAL TRIAL: NCT05477953
Title: Observational Pregnancy Safety Study of Women Exposed to Nifurtimox During Pregnancy to Describe the Risk of Pregnancy and Maternal Complications and Other Events of Interest on the Developing Fetus, Neonate, and Infant
Brief Title: An Observational Pregnancy Safety Study in Women Who Were Exposed to the Drug Nifurtimox During Pregnancy to Learn About the Risk of Pregnancy Complications and About the Mother's and Baby's Health
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21944
Record Dates: First submitted 2022-05-19; First posted 2022-07-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — Nifurtimox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women exposed to nifurtimox: The study will examine the effects of nifurtimox on fetuses, neonates and infants through 12 months of age who were exposed to nifurtimox in utero and maternal complications of pregnancy in women who were exposed to at least one dose of nifurtimox during pregnancy.
  Interventions: Drug: Nifurtimox (BAYA2502)

INTERVENTIONS:
Drug: Nifurtimox (BAYA2502) — At least 1 dose of nifurtimox

SUMMARY:
This is an observational study in which data from women with Chagas disease who will take or have already taken nifurtimox during pregnancy and the impact on their babies are studied.

Chagas disease is an inflammatory, infectious disease caused by the parasite Trypanosoma cruzi. This parasite is mainly spread by insects called triatomine bug. If Chagas disease is left untreated, it can later cause e.g. serious heart and digestive problems.

Nifurtimox has been used for more than 50 years to treat Chagas disease in children and adults.

It is not recommended to be used during pregnancy as data from animal studies indicate that it may harm the baby. Currently, there are not enough data to know if this is also the case in humans.

In this study, researchers want to collect data on the safety of nifurtimox use in pregnant women. To do this, researchers will collect the following information:

* Birth defects (abnormal and problematic structures or functions, a child is born with)
* Pregnancy outcomes (like live birth, preterm birth, still birth/death of the unborn baby, miscarriage, or abortion)
* Certain health problems of the child up to 12 months of age
* Certain health problems of the women experienced during pregnancy The data will be collected from different sources including telephone calls with the women or their doctor, CRFs (case reprt forms) or from medical records The researchers will compare the proportion of children with birth defects, pregnancy outcomes or certain health problems of the child or the women during pregnancy with available data on these outcomes in the general population.

The study will run for approximately 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Females exposed to at least 1 dose of nifurtimox at any time during pregnancy (i.e., from the first day of the last menstrual period / time of conception to pregnancy outcome).
* Written informed consent (for adolescents under the age of majority, written informed assent by the pregnant minor (where applicable) and written informed consent by the parent/legal guardian).

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will actively pursue and attempt to capture all nifurtimox exposures during pregnancy that occur in all countries where nifurtimox is approved to be marketed by Bayer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2032-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Major Congenital Malformations (birth defects) | Up to pregnancy week 40
  1. any major structural defect diagnosed with signs/symptoms, using the selected major congenital anomalies list extracted from the Birth defects surveillance: a manual, CDC.
  2. on a case-by-case basis, through evaluator review and agreement from external advisors (if required), any structural defect (that satisfy criterion 1 or 2) detected in the prenatal evaluation of a pregnancy or in the gross or pathologic examination of an abortus, fetus, or deceased infant will be included, if available, to increase the sensitivity of pregnancy study monitoring

SECONDARY OUTCOMES:
Events of Interest in Neonates and Infants through 12 Months of Age: Hospitalizations for serious illness | Up to 12 months of age
Events of Interest in Neonates and Infants through 12 Months of Age: Medications | Up to 12 months of age
Events of Interest in Neonates and Infants through 12 Months of Age: Growth and development milestones | Up to 12 months of age
  Apgar Scale, CDC Growth Calculators, Cognitive Checklists, ASD (autism spectrum disorder) Tool
Events of Interest in Neonates and Infants through 12 Months of Age: Neonatal or infant mortality | Up to 12 months of age
Maternal Complications: Premature rupture of membranes (PROM) | Up to pregnancy week 40
Maternal Complications: Preeclampsia | Up to pregnancy week 40
Maternal Complications: Severe pregnancy-induced hypertension (PIH) | Up to pregnancy week 40
Maternal Complications: Proteinuria | Up to pregnancy week 40
Maternal Complications: Gestational diabetes | Up to pregnancy week 40
Maternal Complications: Measures of fetal growth deficiency (small for gestational age) | Up to pregnancy week 40
Spontaneous abortion | Up to 20 weeks
  Any loss of a fetus due to natural causes less than 20 weeks gestation as a spontaneous abortion (WHO/CDC/ICBDSR, 2014). If available, data from gross or pathological examination of the abortus or fetus will be evaluated for structural defects.
Elective/Induced abortion | Up to pregnancy week 40
  Elective or induced abortion is the termination of pregnancy through medical or surgical procedures (ACOG, 2014) (WHO, 2014) If available, data from gross or pathological examination of the abortus or fetus will be evaluated for structural defects.
Fetal death/Still birth | More than 20 weeks gestation or weighing less than 500 grams
  Fetal death or stillbirth refers to fetuses born dead at > 20 weeks gestation or weighing > 500 grams.
  Fetal death occurring > 20 weeks but less than 28 weeks gestation is considered an early fetal loss.
  Fetal death occurring > 28 weeks is considered a late fetal loss (ACOG, 2014). If available, data from gross or pathological examination of the abortus or fetus will be evaluated for structural defects.
  • The study will make the final classification between fetal death/still birth and spontaneous abortion based on gestational age and weight. If these parameters are not available, the study will accept the classification indicated by the HCP.
Preterm delivery | Prior to 37 completed weeks of gestation
  Births delivered prior to 37 completed weeks of gestation per 100 births. Gestational age is based on the obstetric estimate of gestation (CDC).
Live Birth | Up to pregnancy week 40
  A live birth refers to a complete expulsion from its mother of a surviving neonate breathing or showing any evidence of life such as a heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles, whether the umbilical cord has been cut or the placenta is attached (WHO, 2014).
Ectopic or Molar Pregnancy | Up to pregnancy week 40
  Any reported ectopic or molar pregnancy will be sub-classified in the respective pregnancy outcome including induced abortion, live birth, or spontaneous pregnancy loss. CDC National Center for Health Statistics surveillance system (NCHS, 2004 ).

CONTACTS AND LOCATIONS:
Locations (11):
- Many Locations, Multiple Locations, West Virginia, United States
- Many Locations, Multiple Locations, Argentina
- Many Locations, Multiple Locations, Bolivia
- Many Locations, Multiple Locations, Chile
- Many Locations, Multiple Locations, El Salvador
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Guatemala
- Many locations, Multiple Locations, Honduras
- Many Locations, Multiple Locations, Mexico
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Uruguay

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com